CLINICAL TRIAL: NCT05607446
Title: A Single-center, Randomized, Double-blind, Two-cycle, Two-way Crossover Phase Ib Study to Evaluate the Efficacy and Safety of TQC3564 Tablets in the Treatment of Persistent Allergic Rhinitis
Brief Title: To Evaluate the Efficacy and Safety of TQC3564 Tablets in the Treatment of Persistent Allergic Rhinitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was closed per sponsor request. Premature closure was not prompted by any safety or efficacy concerns.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC3564-Ib-02
Record Dates: First submitted 2022-10-16; First posted 2022-11-07 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TQC3564 tablets (Experimental): Orally administer TQC3564 tablets for 14 days.
  Interventions: Drug: TQC3564 tablets
- placebo tablets (Placebo Comparator): Orally administer placebo tablets for 14 days.
  Interventions: Drug: Placebo tablets
- TQC3564 tablets + montelukast sodium tablets (Experimental): Orally administer TQC3546 tablets combined with Montelukast sodium tablets for 14 days.
  Interventions: Drug: TQC3564 tablets, montelukast sodium tablets
- placebo tablets + montelukast sodium tablets (Placebo Comparator): Orally administer placebo tablets combined with Montelukast sodium tablets for 14 days.
  Interventions: Drug: Placebo tablets, montelukast sodium tablets

INTERVENTIONS:
Drug: TQC3564 tablets — TQC3564 tablets are CRTH2 antagonists.
  Arms: TQC3564 tablets
Drug: Placebo tablets — The intervention drug is placebo.
  Arms: placebo tablets
Drug: TQC3564 tablets, montelukast sodium tablets — The intervention drugs are TQC3564 tablets combined with montelukast sodium tablets. TQC3564 is a CRTH2 antagonist, montelukast sodium is Leukotriene receptor antagonist.
  Arms: TQC3564 tablets + montelukast sodium tablets
Drug: Placebo tablets, montelukast sodium tablets — The intervention drugs are placebo combined with montelukast sodium tablets. Montelukast sodium is Leukotriene receptor antagonist.
  Arms: placebo tablets + montelukast sodium tablets

SUMMARY:
A clinical study to evaluate the efficacy and safety of tqc3564 tablets in the treatment of persistent allergic rhinitis. A total of 24 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~65 years old, male or female;
* Meet the clinical diagnostic criteria for allergic rhinitis, and the diagnosis is based on the "Guidelines for the Diagnosis and Treatment of Allergic Rhinitis (2015, Tianjin)" issued by the Rhinology Group of the Otolaryngology Head and Neck Surgery Branch of the Chinese Medical Association:

  1. Symptoms: sneezing 2 or more symptoms, such as watery mucus, nasal itching and nasal congestion, persist or accumulate for more than 1 hour per day, and may be accompanied by eye symptoms such as itching, watering and redness;
  2. Signs: Pale and edema of the nasal mucosa is common. Nasal watery secretions;
  3. Allergen test: at least one allergen SPT and/or serum-specific IgE positive (test results within 12 months before screening);
* Female subjects of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; negative serum pregnancy test within 14 days before study enrollment , and must be non-lactating subjects; male subjects should agree to use contraception during the study period and for 6 months after the end of the study period.
* The subjects voluntarily joined the study, signed the informed consent, and had good compliance.

Exclusion Criteria:

* Patients with non-allergic rhinitis, such as drug-induced rhinitis, vasomotor rhinitis, non-allergic rhinitis eosinophilic rhinitis, etc.; patients with severe nasal septum deviation, sinusitis, nasal polyps, hypertrophic rhinitis Other nasal organic lesions;
* In the nasal examination at the end of the screening period or the introduction period, there is any erosion of the nasal mucosa, septal ulcer or perforation of the nasal septum;
* Those who have undergone sinus surgery within 3 months before the screening period or who have not fully healed the nasal wound;
* The subject has uncontrolled diabetes mellitus, that is, fasting blood glucose (FBG) > 10mmol/L in the laboratory test during the screening period;
* History of allergy to any study drug or similar chemical drugs (CRTh2 antagonists);
* History of severe allergic reaction to any allergen, such as anaphylactic shock or life-threatening asthma, previous intubation, respiratory arrest, hospitalization for asthma or acute asthma attack within the past 3 months;
* Those who were found to respond to placebo during the lead-in period (with rhinitis symptoms of moderate or above during the screening period, those with mild or no symptoms during the lead-in period, or baseline rTNSS mean <6 points were defined as placebo responders;
* Women who are pregnant or breastfeeding, or who plan to become pregnant or breastfeeding during the study period;
* Any subject deemed unsuitable for participation in this clinical study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Total nasal symptom Score (TNSS) | Baseline, Day 14
  Change in the investigator-assessed total nasal symptom score (TNSS) from baseline to 14 days. TNSS was the sum score of 4 nasal symptoms with a minimum score of 0 units and a maximum score of 12 units, with higher score corresponding to increased nasal allergy symptoms.

SECONDARY OUTCOMES:
Total ocular symptom score(TOSS) | Baseline, Day 14
  Change in the TOSS from baseline to14 days. TOSS was the sum of 2 ocular symptoms with a minimum score of 0 units and amaximum score of 6 units, with higher score corresponding to increased ocular symptoms.
Individual Total Nasal Symptom Score (TNSS) | Baseline, Day 14
  Change in the individual TNSS from baseline to 14 days. Individual nasal symptoms were each rated on a 4-point scale from 0-3 (0=Absent, 1=Mild, 2=Moderate, 3=Severe), with no half-unit assessments.
Individual Total Ocular Symptom Score (TOSS) | Baseline, Day 14
  Change in the individual TOSS from baseline to 14 days. Individual ocular symptoms were each rated on a 4-point scale from 0-3 (0=Absent, 1=Mild, 2=Moderate, 3=Severe), with no half-unit assessments.
Daily symptoms score (dSS) | Baseline, Day 14
  Change in the dSS from baseline to 14 days. dSS was the sum of 4 nasal symptoms and 2 ocular symptoms with a minimum score of 0 units and amaximum score of 18 units, with higher score corresponding to increased overall symptoms.
Rescue medication proportion | Day 1-32
  Proportion of participants using rescue medication mometasone furoate nasal spray during intervention
Rescue medication frequency | Day 1-32
  Frequency of using rescue medication mometasone furoate nasal spray during intervention
Incidence of adverse events | Day 1-32
  Incidence of adverse events, including vital signs, physical examination, abnormal laboratory parameters, etc.,

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No